CLINICAL TRIAL: NCT05573503
Title: Effects of a Web Based Education Programme About Sexuality Aimed at Nurses That Care for Patients With Cancer (Sex-Can WebEd Nurse)
Brief Title: Effects of a Web Based Education Programme About Sexuality Aimed at Nurses That Care for Patients With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karlstad University (Other)
Responsible Party: Principal Investigator, Cecilia Olsson, PhD, Senior lecturer, associate professor, Karlstad University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SexCanWebEdNurse
Record Dates: First submitted 2022-10-03; First posted 2022-10-10 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Neoplasms; Nurse-Patient Relations; Sexuality
Keywords: web based education; cancer nurses
MeSH Terms: conditions — Neoplasms; Sexuality | interventions — Oncology Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants complete baseline assessments and are then assigned the intervention.
  Interventions: Other: Bring it up - Assessment and support of patients' sexuality in cancer nursing

INTERVENTIONS:
Other: Bring it up - Assessment and support of patients' sexuality in cancer nursing — Participants will attend a five week online university course, "Bring it up - Assessment and support of patients' sexuality in cancer nursing". The course addresses theories and models about sexuality in relation to cancer illness, conversation techniques, models for addressing sensitive topics, methods for assessing the impact of cancer on sexuality, methods for preventing and treating sexual problems in relation to cancer, relevant nursing interventions for person-centred counselling about sexuality, and ethical aspects.
  The teaching consists of literature, online lectures, seminars, clinical practice, and written exams. A university certificate will be issued to participants who pass all exams.

SUMMARY:
The purpose of the SexCan - WebEd Nurse study is to evaluate the effect of a five week online university course, "Bring it up - Assessment and support of patients' sexuality in cancer nursing", aimed at cancer nurses, on occupational self-efficacy and attitudes towards addressing sexuality with patients.

DETAILED DESCRIPTION:
Cancer nurses attending the course will be recruited. Effects will be used with a pre-post design at two occasions or until we reach 15 participants. Survey data will be collected at baseline and two times post the course. Qualitative interviews with participants will also be performed as well as observational data from the seminars in the course.

The participants' ward managers will also be invited to qualitative interviews considering how to implement the nurses' new knowledge clinically.

ELIGIBILITY:
Inclusion Criteria:

- Registered nurses working as a contact nurses in cancer care who are admitted to the intervention university course.

Exclusion Criteria:

- N/A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Occupational Self-Efficacy (from baseline to 5 weeks post finished intervention) | At baseline and then 5 weeks post finished intervention.
  Measured with the "Short Occupational Self-Efficacy Scale". This instrument ranges from 6 to 36 points, where higher values indicate a higher grade of self-efficacy.
Change in Occupational Self-Efficacy (from baseline to 19 weeks post finished intervention) | At baseline and then 19 weeks post finished intervention.
  Measured with the "Short Occupational Self-Efficacy Scale"
Change in Attitudes towards addressing sexuality (from baseline to 5 weeks post finished intervention) | At baseline and then 5 weeks post finished intervention.
  Measured with the "Sexual Health - Extended Version - Swedish (PASH-Ext-S)". The instrument ranges from 27 to 135 points. Higher values indicate a higher degree of positive attitudes to addressing sexuality.
Change in Attitudes towards addressing sexuality (from baseline to 19 weeks post finished intervention) | At baseline and then 19 weeks post finished intervention.
  Measured with the "Sexual Health - Extended Version - Swedish (PASH-Ext-S)"

SECONDARY OUTCOMES:
Change in Knowledge about the influence of cancer on sexuality (from baseline to 5 weeks post finished intervention) | At baseline and then 5 post finished intervention.
  Study specific questionnaire
Change in Knowledge about the influence of cancer on sexuality (from baseline to 19 weeks post finished intervention) | At baseline and then 19 weeks post finished intervention.
  Study specific questionnaire
Change in Number of conversations with patients relating to sexuality (from baseline to 5 weeks post finished intervention) | At baseline and then 5 weeks post finished intervention.
Change in Number of conversations with patients relating to sexuality (from baseline to 5 weeks post finished intervention) | At baseline and then 19 weeks post finished intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Olsson, PhD, Principal Investigator — Karlstad University
Locations (1):
- Karlstad University, Karlstad, Värmland County, Sweden